CLINICAL TRIAL: NCT03720691
Title: Effect of Repetitive Transcranial Magnetic Stimulation in Vascular Parkinsonism
Brief Title: rTMS Treatment in Vascular Parkinsonism
Acronym: rTMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Inje University (Other)
Collaborators: Dongtan Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Sangjin Kim, Professor, Inje University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18-0089
Record Dates: First submitted 2018-10-22; First posted 2018-10-25 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Vascular Parkinsonism
Keywords: parkinsonism; vascular parkinsonism; repetitive transcranial magnetic stimulation; brain stimulation
MeSH Terms: conditions — Parkinsonian Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real rTMS Supplementary motor area (Active Comparator): Real rTMS will be applied over the supplementary motor area
  Interventions: Device: Real rTMS Supplementary motor area
- Sham rTMS Supplementary motor area (Sham Comparator): Sham rTMS will be applied over the supplementary motor area
  Interventions: Device: Sham rTMS Supplementary motor area

INTERVENTIONS:
Device: Real rTMS Supplementary motor area — There will be a series of four rTMS blocks separated by 10 minutes. Each block will consist of 15 to 25 pulse trains of 1-second duration at 25 Hz, with an intertrain interval of 10 seconds.
  Other Names: Real repetitive transcranial magnetic stimulation
  Arms: Real rTMS Supplementary motor area
Device: Sham rTMS Supplementary motor area — There will be no real brain stimulation in Sham rTMS, and participant will be blinded.
  Other Names: Sham repetitive transcranial magnetic stimulation
  Arms: Sham rTMS Supplementary motor area

SUMMARY:
Vascular parkinsonism (VP), parkinsonism resulting from ischemic cerebrovascular disease, was suggested in 1929. The main features are wide-based gait, postural instability, and falls, which make patients with VP frustrated. Currently, the treatment is challenging.

Transcranial magnetic stiumation is a noninvasive procedure using electromagnetic induction to stimulate brain, and repetitive transcranial magnetic stiumation (rTMS) can selectively change brain activity to enhance desired effects. The aim of this study is to explore the therapeutic effect of rTMS for the VP.

ELIGIBILITY:
Inclusion Criteria:

* Vascular parkinsonism
* age 18 and older

Exclusion Criteria:

* pregnant or any, other medical, surgical, neurological or psychiatric conditions
* other restrictions which prevent you from undergoing TMS recording, such as; surgically or traumatically implanted foreign bodies such as a pacemaker, an implanted medication pump, a metal plate in the skull, or metal inside the skull or eyes (other than dental appliances or fillings), and/ or heart/cardiac lines
* any past or current history of seizure disorder or epilepsy
* unable to give informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (UPDRS) part III-motor part (Number 18 ~31 of UPDRS) | 2 days
  Motor functions will be checked using UPDRS. Each item of the motor part ranges from 0 to 4 (0 means normal, 4 means worst condition). Total sum will be calculated.

SECONDARY OUTCOMES:
Finger tapping test with right hand | 2 days
  Finger tapping test with right hand, as quickly as possible for 15 second. The total number of taps will be calculated. The test will be twice with one minute interval. After the test performed twice, the average of the tests will be used.
The total number of steps during the stand-walk-sit (SWS) test | 2 days
  SWS test is Standing up, making a 9 m round trip, and sitting down as quickly as possible. The number of steps will be recorded.
The completion time during the SWS test | 2 days
  The completion time will be recorded.
Freezing episodes of gait trajectory | 2 days
  The number of freezing episodes during rapid full turns and dual task
Patient and Clinical Global Impression Scale | 2 days
  7-point scale that requires the patient (or clinician) to rate the response of the interventions. The rating will be numbered (1: very much improved; 2: much improved; 3: minimally improved; 4: no changes; 5: minimally worse; 6: much worse; 7: very much worse).

CONTACTS AND LOCATIONS:
Overall Officials: Sang Jin Kim, MD, PhD, Principal Investigator — Inje Unversity, Busan Paik Hospital
Locations (1):
- Inje university, Busan Paik Hospital, Busan, South Korea